CLINICAL TRIAL: NCT03257267
Title: An Open-Label, Randomized, Phase 3 Clinical Trial of REGN2810 Versus Investigator's Choice of Chemotherapy in Recurrent or Metastatic Cervical Carcinoma
Brief Title: Study of Cemiplimab in Adults With Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1676; 2017-000350-19 (EudraCT Number)
Record Dates: First submitted 2017-07-26; First posted 2017-08-22 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Squamous Cell Carcinoma (SCC); Recurrent or Metastatic, Platinum-refractory Cervical Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Recurrence; Neoplasm Metastasis | interventions — cemiplimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Therapy (Experimental): Cemiplimab
  Interventions: Drug: Cemiplimab
- Control Therapy (Active Comparator): Investigator choice (IC) chemotherapy
  Interventions: Drug: Investigator Choice (IC) Chemotherapy

INTERVENTIONS:
Drug: Cemiplimab — Intravenous (IV) administration every 3 weeks (Q3W)
  Other Names: REGN2810; Libtayo
  Arms: Experimental Therapy
Drug: Investigator Choice (IC) Chemotherapy — IC chemotherapy options include:
  1. Antifolate: Pemetrexed
  2. Topoisomerase 1 inhibitor: Topotecan or Irinotecan
  3. Nucleoside analogue: Gemcitabine
  4. Vinca alkaloid: Vinorelbine
  The only chemotherapy treatments allowed in the control arm are any of the 5 drugs that are listed as IC options above.
  Arms: Control Therapy

SUMMARY:
The primary objective is to compare overall survival (OS) for patients with recurrent or metastatic cervical cancer who have histology of squamous cell carcinoma (SCC) and who have any eligible histology treated with either cemiplimab or investigator's choice (IC) chemotherapy.

The secondary objectives performed among SCC patients and among all eligible histologies (SCC and adenocarcinoma/adenosquamous carcinoma (AC) are:

* To compare progression-free survival (PFS) of cemiplimab versus IC chemotherapy
* To compare objective response rate (ORR) (partial response [PR] + complete response [CR]) of cemiplimab versus IC chemotherapy per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* To compare the duration of response (DOR) of cemiplimab versus IC chemotherapy
* To compare the safety profiles of cemiplimab versus IC chemotherapy by describing adverse events (AE)
* To compare quality of life (QOL) for patients treated with cemiplimab versus IC chemotherapy using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30)

ELIGIBILITY:
The criteria listed below are not intended to contain all considerations relevant to a patient's potential participation in this clinical trial.

Key Inclusion Criteria:

1. Recurrent, persistent, and/or metastatic cervical cancer with squamous cell histology, for which there is not a curative-intent option (surgery or radiation therapy with or without chemotherapy).

   * Acceptable histologies (squamous carcinoma, adenocarcinoma, and adenosquamous carcinoma) as defined in the protocol
2. Tumor progression or recurrence after treatment with platinum therapy (must have been used to treat metastatic, persistent, or recurrent cervical cancer)
3. Patient must have measurable disease as defined by RECIST 1.1.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
5. ≥18 years old
6. Adequate organ or bone marrow function
7. Received prior bevacizumab therapy or had clinically documented reason why not administered
8. Received prior paclitaxel therapy or had clinically documented reason why not administered

Key Exclusion Criteria:

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments
2. Prior treatment with an agent that blocks the PD-1/PD-L1 pathway
3. Prior treatment with other systemic immune-modulating agents that was

   1. within fewer than 4 weeks (28 days) of the enrollment date, or
   2. associated with irAEs of any grade within 90 days prior to enrollment, or
   3. associated with toxicity that resulted in discontinuation of the immune modulating agent
4. Active or untreated brain metastases
5. Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of study drug cemiplimab or IC chemo)
6. Active infection requiring therapy
7. History of pneumonitis within the last 5 years
8. History of documented allergic reactions or acute hypersensitivity reaction attributed to antibody treatments
9. Concurrent malignancy other than cervical cancer and/or history of malignancy other than cervical cancer within 3 years of date of first planned dose of study drug cemiplimab or IC chemo), except for tumors with negligible risk of metastasis or death, such as adequately treated cutaneous squamous cell carcinoma or basal cell carcinoma of the skin or ductal carcinoma in situ of the breast. Patients with hematologic malignancies (eg, chronic lymphocytic leukemia) are excluded.

Note: Other protocol defined Inclusion/Exclusion apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (105):
- United States (11):
  - Arizona Oncology Associates, Phoenix, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - University of California Irvine, Orange, California
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Cancer Research for the Ozarks, Springfield, Missouri
  - New York Presbyterian Queens, Flushing, New York
  - Northwell Health, Lake Success, New York
  - Laura and Issac Perlmutter Cancer Center at NYU Langone, New York, New York
  - First Health of the Carolinas Outpatient Cancer Center, Pinehurst, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Texas Oncology, P.A., Austin, Texas
- Australia (6):
  - St. George Hospital, Kogarah, New South Wales
  - Northern NSW Health District, The Tweed Hospital, Tweed Heads, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St. John of God Subiaco Hospital, Subiaco, Western Australia
- Belgium (7):
  - OLV ziekenhuis Aalst, Medische oncologie- Radiotherapie, Aalst
  - Institut Bordet, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - UZLeuven Gynaelologic Oncology, Leuven
  - CHC Saint Joseph, Liège
  - CHU Liège, Liège
  - CHU UCL Namur site Sainte Elisabeth, Namur
- Brazil (8):
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Hosptial Sao Lucas da PUC de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Novos Tratamentos Itajai, Itajaí, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Instituto de Pesquisas Clinicas para Estudos Multicentricos - IPCEM, Caxias do Sul
  - Instituto Nacional de Cancer - INCA, Rio de Janeiro
  - Instituto COI de Pesquisa, Rio de Janeiro
- Canada (7):
  - Tom Baker Cancer Center, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Hopital Notre-Dame du Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Greece (4):
  - General Hospital of Athens Alexandra, Athens
  - University Hospital of Ioannina, Ioannina
  - General Hospital of Patras, Pátrai
  - Euromedica General Clinic, B'Oncology Clinic, Thessaloniki
- Italy (8):
  - Azienda Ospedaliero Universitaria di Bologna, Bologna
  - U.O Oncologia Medica P.O Vito Fazzi, Lecce
  - Asst Lecco, Lecco
  - Irst Irccs, Meldola
  - Istituto Europeo di Oncologia, Milan
  - AUSL, IRCCS di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Agostino Gemelli IRCCS di Roma, Roma
  - Regina Elena National Cancer Institute, Rome
- Japan (14):
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - Fukui University Hospital, Yoshida-gun, Fukui
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa
  - Saitama Medical University, Saitama, Saitama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Saitama Cancer Center, Saitama, Tokyo
  - National Kyushu Cancer Center, Fukuoka
  - Kagoshima City Hospital, Kagoshima
- Poland (5):
  - Bialostockie Centrum Onkologii, Bialystok
  - Szpitale Pomorskie, Gdynia
  - Center and Institute of Oncology Gliwice, Gliwice
  - Centrum Onkologii Ziemi Lubelskiej im sw. Jana z Dukli, Lublin
  - Greater Poland Cancer Center, Poznan
- Russia (9):
  - Regional Budgetary Institution of Healthcare Ivanovo Regional Oncology Dispensary, Ivanovo, Ivanovo Oblast
  - State Budgetary Healthcare Institution "Oncology Dispensary" of Ministry of Healthcare of the Kabardino-Balkarian Republic, Nal'chik, Kabardino-Balkarian
  - A. Tsyb Medical Radiological Research Center, Obninsk, Kaluga Oblast
  - State Budgetary Institution of Healthcare, Clinical Oncology Dispensary #1 of Ministry of Health of Krasnodar Region, Krasnodar, Krasnodar Territory
  - State Budgetary Healthcare Institution Leningrad Regional Oncological Dispensary (SBHI "LROD"), Vsevolozhsk, Leningradskaya Oblast'
  - State Autonomous Healthcare Institution ,Republican Clinical Oncological Dispensary of the Ministry of Healthcare of the Tatarstan Republic, Kazan', Tatarstan Republic
  - Budgetary Institution of Healthcare of Omsk region Clinical Oncology Dispensary, Omsk
  - State Budgetary Institution of Healthcare "Orenburg Regional Clinical Oncology Dispensary", Orenburg
  - Saint- Petersburg State Budgetary institution of Healthcare "City Clinical Oncological Dispensary", Saint Petersburg
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (10):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Vall d´Hebron University Hospital, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Instituto Catalan de Oncologia de Gerona, Girona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario HM Sanchinarro CIOCC, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - MacKay Memorial Hospital, Taipei
  - Koo-Foundation Sun Yat-Sen Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (6):
  - Velindre Cancer Centre, Cardiff
  - NHS Greater Glasgow and Clyde Beatson, West of Scotland Cancer care, Glasgow
  - University College Hospital, London
  - Royal Marsden NHS Foundation Trust, Chelsea, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Marsden NHS Foundation Trust, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Oaknin A, Monk BJ, Vergote I, Cristina de Melo A, Kim YM, Lisyanskaya AS, Samouelian V, Kim HS, Gotovkin EA, Damian F, Chang CL, Takahashi S, Li J, Mathias M, Fury MG, Ivanescu C, Reaney M, LaFontaine PR, Lowy I, Harnett J, Chen CI, Tewari KS. EMPOWER CERVICAL-1: Effects of cemiplimab versus chemotherapy on patient-reported quality of life, functioning and symptoms among women with recurrent cervical cancer. Eur J Cancer. 2022 Oct;174:299-309. doi: 10.1016/j.ejca.2022.03.016. Epub 2022 Jul 31. PMID 35922251
- [Derived] Tewari KS, Monk BJ, Vergote I, Miller A, de Melo AC, Kim HS, Kim YM, Lisyanskaya A, Samouelian V, Lorusso D, Damian F, Chang CL, Gotovkin EA, Takahashi S, Ramone D, Pikiel J, Mackowiak-Matejczyk B, Guerra Alia EM, Colombo N, Makarova Y, Rischin D, Lheureux S, Hasegawa K, Fujiwara K, Li J, Jamil S, Jankovic V, Chen CI, Seebach F, Weinreich DM, Yancopoulos GD, Lowy I, Mathias M, Fury MG, Oaknin A; Investigators for GOG Protocol 3016 and ENGOT Protocol En-Cx9. Survival with Cemiplimab in Recurrent Cervical Cancer. N Engl J Med. 2022 Feb 10;386(6):544-555. doi: 10.1056/NEJMoa2112187. PMID 35139273
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 752 participants were screened, 144 participants failed screening, 608 participants randomized to receive cemiplimab or investigator choice of chemotherapy. Control treatment determined before randomization by investigator from options per protocol.
Groups:
- Cemiplimab: Participants received a fixed dose of 350 milligrams (mg) of cemiplimab intravenous (IV) infusion on Day 1 of every 3 weeks (Q3W) for up to 96 weeks (up to 16 cycles of 6 weeks each) or until progression of disease or unacceptable toxicity, voluntary withdrawal from the study.
- Investigator Choice (IC) Chemotherapy: Participants received IC of chemotherapy (options listed by class): (1) Antifolate: pemetrexed 500 mg per meter square (mg/m^2) on Day 1; (2) Topoisomerase 1 inhibitor: topotecan 1 mg/m^2 daily for 5 days, starting on Day 1 or irinotecan 100 mg/m^2 weekly (Days 1, 8, 15 and 22), followed by 10 to 14 days rest, for a 42-day (6-week) cycle; (3) Nucleoside analogue: gemcitabine 1000 mg/m^2 on Days 1 and 8; (4) Vinca alkaloid: vinorelbine 30 mg/m^2 IV infusion based on body surface area for Q3W up to 96 weeks (up to 16 cycles of 6 weeks each) or until progression of disease or unacceptable toxicity, voluntary withdrawal from the study.
Period: Overall Study
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Started | 304 | 304
Full Analysis Set (FAS) (The FAS included all randomized participants.) | 304 | 304
Safety Analysis Set (SAF) (The SAF included all randomized participants who received any study drug.) | 300 | 290
Completed Treatment | 38 | 0
Completed (Completed Study) | 35 | 0
Not Completed | 269 | 304
Not completed — Adverse Event | 17 | 7
Not completed — Death | 96 | 98
Not completed — Lost to Follow-up | 2 | 2
Not completed — Non-compliance with Study Drug | 0 | 2
Not completed — Participant Decision | 35 | 43
Not completed — Sponsor Decision | 1 | 0
Not completed — Physician Decision | 1 | 3
Not completed — Disease Progression | 109 | 121
Not completed — Withdrawal by Subject | 8 | 26
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: The FAS included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy | Total
Number analyzed (Participants) | 304 | 304 | 608
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (11.59) | 51.2 (11.77) | 51.1 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 304 | 608
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 44 | 91
  Not Hispanic or Latino | 251 | 250 | 501
  Unknown or Not Reported | 6 | 10 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 193 | 192 | 385
  Black or African American | 9 | 12 | 21
  Asian | 88 | 88 | 176
  American Indian or Alaska Native | 2 | 1 | 3
  Other | 8 | 4 | 12
  Unknown | 1 | 1 | 2
  Not Reported | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to the date of death due to any cause. A participant who had not died was censored at the last known date of contact.
Time Frame: From first dose up to 90 following last dose (~42 months)
Population: The full analysis set (FAS) included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Number analyzed (Participants) | 304 | 304
Months | 11.7 [9.6 to 13.4] | 8.5 [7.5 to 9.6]
Statistical Analysis 1: Comparison: Cemiplimab vs Investigator Choice (IC) Chemotherapy; Test type: Superiority; p < 0.00001, Stratified Log-rank Test — One-sided p-value; Hazard Ratio (HR) = 0.665, 95% CI 2-sided [0.555 to 0.796]

2. Secondary Outcome: Progression-free Survival (PFS) Assessed by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: PFS was defined as the time from randomization to the date of the first documented tumor progression (radiographic) or death due to any cause. Participants who did not have a documented tumor progression or death were censored on the date of their last evaluable tumor assessment.
Time Frame: Time from randomization to the date of the first documented tumor progression or death due to any cause (assessed up to 40 months)
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Number analyzed (Participants) | 304 | 304
Months | 2.8 [2.6 to 3.9] | 2.9 [2.7 to 3.5]
Statistical Analysis 1: Comparison: Cemiplimab vs Investigator Choice (IC) Chemotherapy; Test type: Superiority; p = 0.00031, Stratified Log-rank Test; Hazard Ratio (HR) = 0.741, 95% CI 2-sided [0.623 to 0.882]

3. Secondary Outcome: Objective Response Rate (ORR) Assessed by Investigator Using RECIST 1.1
Description: ORR was defined as the number of participants who achieved complete response (CR) or partial response (PR) as per RECIST 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm) (<1 centimeter [cm]). PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization up to 40 months
Population: The FAS included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Number analyzed (Participants) | 304 | 304
Participants | 52 | 19
Statistical Analysis 1: Comparison: Cemiplimab vs Investigator Choice (IC) Chemotherapy; Test type: Superiority; p = 0.00002, Stratified Cochran-Mantel-Haenszel test; Odds Ratio (OR) = 3.136, 95% CI 2-sided [1.798 to 5.468]

4. Secondary Outcome: Duration of Response (DOR) Assessed Per RECIST 1.1
Description: DOR was defined as the time from the date of first response (CR or PR) to the date of the first documented progressive disease (per RECIST 1.1) or death due to any cause. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm). PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Participants who never progressed while being followed was censored at the last valid tumor measurement. DOR was determined by Kaplan-Meier estimate.
Time Frame: Time from the date of first response to the date of the first documented progressive disease or death due to any cause (up to 40 months)
Population: The FAS included all randomized participants with confirmed CR or PR. Here 'n' = number of evaluable participants at a specified timeframe.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Number analyzed (Participants) | 52 | 19
Months | 18.7 [16.4 to NA] — Insufficient number of participants with events | 7.2 [5.1 to 9.9]

5. Secondary Outcome: Quality of Life (QoL): Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) of Global Health Status /Quality of Life (GHS/QoL) and Physical Functioning Scales
Description: EORTC QLQ-C30 is a 30-question tool used to assess the overall QoL in cancer participants. It consisted of 15 domains: 1 GHS/QoL scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact). Most items are scored 1 ("not at all") to 4 ("very much") except for the items contributing to the GHS/QoL, which are scored 1 ("very poor") to 7 ("excellent"). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100. For the GHS/QoL and 5 functional scales a high score indicates better global health status/functioning and a negative change from baseline indicated less improvement. For the symptom scales, a high score indicates a higher level of symptoms, and a negative change from baseline indicated an improvement in symptoms.
Time Frame: From Cycle 1 Day 1 up to 40 months (Each cycle = 42 days)
Population: The FAS included all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Number analyzed (Participants) | 304 | 304
Score on a Scale
  Overall: Change from Baseline of EORTC QLQ-C30 GHS/QoL | 0.46 [-2.715 to 3.642] | -8.54 [-13.004 to -4.084]
  Overall: Changes from Baseline of EORTC QLQ-C30 Physical Functioning | -0.27 [-3.014 to 2.473] | -8.86 [-12.517 to -5.196]

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Death
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. A Treatment-emergent adverse event (TEAE) was defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life- threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious TEAEs. Number of participants with TEAEs, serious TEAEs, and TEAEs leading to death were reported.
Time Frame: From first dose up to 90 following last dose (~36 months)
Population: The safety analysis set (SAF) included all randomized participants who received any study drug. Here 'n' = number of evaluable participants at a specified timeframe.
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Number analyzed (Participants) | 300 | 290
Participants
  Participants with any TEAE | 269 | 266
  Participants with any Serious TEAE | 96 | 78
  Participants with any TEAE leading to Death | 5 | 2

7. Secondary Outcome: Number of Participants With New or Worsened Laboratory Results by National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE) Grade
Description: Laboratory parameters included hematology, electrolytes, chemistry (other), and liver function. Clinically significant abnormalities were determined by the investigator based on NCI-CTCAE Grade where Grade 1 = Mild, Grade 2 = moderate, Grade 3 = severe; Grade 4 = life threatening or disabling; Grade 5 = death. Participants with at least 1 lab abnormality Graded 3/4 in hematology, electrolytes, chemistry (other), or liver function reported.
Time Frame: From first dose up to 90 following last dose (~36 months)
Population: The SAF included all randomized participants who received any study drug. Here 'n' = number of evaluable participants at a specified timeframe.
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Number analyzed (Participants) | 300 | 290
Participants
  Hematology (Grades 3/4): number analyzed (Participants) | 293 | 278
  Hematology (Grades 3/4) | 84 | 137
  Electrolytes (Grades 3/4): number analyzed (Participants) | 294 | 271
  Electrolytes (Grades 3/4) | 47 | 32
  Chemistry (Other) (Grades 3/4): number analyzed (Participants) | 294 | 272
  Chemistry (Other) (Grades 3/4) | 12 | 10
  Liver Function (Grades 3/4): number analyzed (Participants) | 294 | 271
  Liver Function (Grades 3/4) | 28 | 23

8. Primary Outcome: Overall Survival (OS) in the SCC Population
Description: as for outcome 1
Time Frame: From first dose up to 90 following last dose (~42 months)
Population: All randomized participants who presented SCC (Squamous cell carcinoma) histology. Here 'n' = the number of evaluable participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cemiplimab | Investigator Choice (IC) Chemotherapy
Number analyzed (Participants) | 239 | 238
Months | 10.9 [8.9 to 12.9] | 8.8 [7.6 to 9.8]
Statistical Analysis 1: Comparison: Cemiplimab vs Investigator Choice (IC) Chemotherapy; Test type: Superiority; p = 0.00024, Stratified Log-rank Test — One-sided p-value; Hazard Ratio (HR) = 0.698, 95% CI 2-sided [0.570 to 0.855]

ADVERSE EVENTS:
Time Frame: From first dose up to 90 following last dose (~42 months)
Groups:
- Chemotherapy*: Participants received IC of chemotherapy (options listed by class): (1) Antifolate: pemetrexed 500 mg per meter square (mg/m^2) on Day 1; (2) Topoisomerase 1 inhibitor: topotecan 1 mg/m^2 daily for 5 days, starting on Day 1 or irinotecan 100 mg/m^2 weekly (Days 1, 8, 15 and 22), followed by 10 to 14 days rest, for a 42-day (6-week) cycle; (3) Nucleoside analogue: gemcitabine 1000 mg/m^2 on Days 1 and 8; (4) Vinca alkaloid: vinorelbine 30 mg/m^2 IV infusion based on body surface area for Q3W up to 96 weeks (up to 16 cycles of 6 weeks each) or until progression of disease or unacceptable toxicity, voluntary withdrawal from the study.
- Chemotherapy to Cemiplimab*: Treatment until disease progression, unacceptable toxicity, or voluntary withdrawal from the study, or until 96 weeks (16 cycles, each 6 weeks). Participants received a fixed dose of 350 milligrams (mg) of cemiplimab intravenous (IV) infusion on Day 1 of every 3 weeks (Q3W) for up to 96 weeks (up to 16 cycles of 6 weeks each) or until progression of disease or unacceptable toxicity, voluntary withdrawal from the study.
Arm/Group | Cemiplimab | Chemotherapy* | Chemotherapy to Cemiplimab*
All-Cause Mortality (participants affected / at risk) | 234/300 | 249/290 | 2/8
Serious Adverse Events (participants affected / at risk) | 100/300 | 84/290 | 1/8
Other Adverse Events (participants affected / at risk) | 239/300 | 253/290 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab (N=300) | Chemotherapy* (N=290) | Chemotherapy to Cemiplimab* (N=8)
Urinary tract infection (Infections and infestations) | 15 (19) | 11 (13) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 3 (4) | 0 (0)
Pyelonephritis (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 1 (4) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Toxic shock syndrome streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (5) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyomyositis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 14 (19) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Oral papule (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 3 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (4) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 6 (7) | 0 (0)
Catheter site thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Device use error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 4 (4) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab (N=300) | Chemotherapy* (N=290) | Chemotherapy to Cemiplimab* (N=8)
Nausea (Gastrointestinal disorders) | 63 (74) | 100 (175) | 0 (0)
Vomiting (Gastrointestinal disorders) | 49 (65) | 66 (101) | 0 (0)
Constipation (Gastrointestinal disorders) | 46 (50) | 58 (64) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 35 (61) | 41 (60) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 28 (31) | 34 (52) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 12 (12) | 22 (24) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 79 (99) | 128 (161) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 9 (11) | 45 (75) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 15 (17) | 0 (0)
Pyrexia (General disorders) | 36 (54) | 62 (117) | 2 (2)
Asthenia (General disorders) | 35 (37) | 45 (63) | 0 (0)
Fatigue (General disorders) | 52 (54) | 45 (81) | 0 (0)
Oedema peripheral (General disorders) | 22 (22) | 16 (16) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (7) | 26 (64) | 0 (0)
Alanine aminotransferase increased (Investigations) | 14 (14) | 20 (26) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 14 (19) | 19 (25) | 0 (0)
Blood creatinine increased (Investigations) | 19 (26) | 16 (16) | 0 (0)
White blood cell count decreased (Investigations) | 2 (3) | 17 (35) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 46 (49) | 46 (55) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 23 (26) | 19 (19) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (23) | 17 (20) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 16 (21) | 0 (0)
Urinary tract infection (Infections and infestations) | 27 (36) | 18 (25) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (37) | 28 (29) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (38) | 8 (11) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (20) | 8 (9) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 19 (29) | 19 (22) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (19) | 15 (15) | 0 (0)
Headache (Nervous system disorders) | 22 (43) | 18 (19) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 21 (28) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 18 (22) | 0 (0)
Insomnia (Psychiatric disorders) | 20 (21) | 17 (18) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 13 (14) | 16 (16) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 15 (16) | 6 (9) | 0 (0)
Hypothyroidism (Endocrine disorders) | 17 (17) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (8) | 13 (38) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 9 (9) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT03257267/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT03257267/SAP_001.pdf